CLINICAL TRIAL: NCT02806063
Title: Bacteriological Setting Before Prosthesis Implantation With One Stage Surgery in Prosthetic Joint Infection
Acronym: Bac-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, SMARMOR, Orthopaedic surgeon, Groupe Hospitalier Diaconesses Croix Saint-Simon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ID RCB : 2015-A01698-41
Record Dates: First submitted 2016-05-25; First posted 2016-06-20 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Prosthetic Joint Infection
Keywords: Prosthesis; joint infection; perioperative samples

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative samples (Other): During this study of health care procedure evaluating microbiological setting in PJI prior prosthesis implantation with one stage surgery, 3 additional perioperative samples will be performed prior prosthesis implantation for every patient.
  Interventions: Procedure: intraoperative samples

INTERVENTIONS:
Procedure: intraoperative samples

SUMMARY:
Chronic prosthetic joint infection (PJI) is a devastating complication of arthroplasty and its treatment continues to fuel the debate on how to manage it appropriately.

One stage and two stage exchange surgery both are the conventional surgical procedures for chronic PJI commonly used to date.

Two stage surgery disadvantages (major surgery, anesthesia and nosocomial risks, functional impairment between surgeries and a high socio-economic coast) encouraged many surgical teams to adopt one stage exchange surgery which provides equivalent or better outcomes. However one stage surgery encounters a major conceptual difficulty when it comes to implant the new prosthesis in a surgical site microbiologically undetermined and potentially contaminated.

Investigators suppose the new prosthesis is implanted in a contaminated setting regardless of bacteria type and antibiotic therapy duration before arthroplasty.

The total lack of data answering this question motivated the conception of this prospective study in order to describe the microbiological setting where is implanted the new prosthesis with one stage exchange surgery after surgical excision and antibiotic therapy initiation in chronic PJI.

DETAILED DESCRIPTION:
Study duration: Two weeks. Recruitment period: 18 months. Maximal duration of data collection: Two weeks. Investigator center: monocenter study. Mean patient inclusion per year: 70 patients per year.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Aged over 18 years
* PJI documented preoperatively by joint fluid culture according to Musculoskeletal Infection Society Definition
* Monoarticular PJI
* PJI management validated at the weekly cross-disciplinary conciliation meeting
* PJI treated with one stage surgery and intravenous antibiotherapy adjusted to preoperative aspiration results.

Exclusion Criteria:

* patient who does not meet eligibility criteria
* Negative preoperative aspiration culture
* PJI du to fungi
* Patient lawfully deprived of his liberty
* Patient insured under social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The number of patients with positive per-operative sample culture after surgical excision and antibiotic initiation and prior prosthesis implantation | 18 months
  In routine care procedure for prosthetic joint infection (PJI), at least, five intraoperative samples are taken before debridement and prosthesis removal in order to identify the causative organism. For the purpose of this study three additional intraoperative samples will be performed after debridement and antibiotic initiation and prior prosthesis implantation.

SECONDARY OUTCOMES:
Description of microbiological evolution of preoperative and perioperative samples before and after surgical excision. | 18 months
  In routine care procedure for prosthetic joint infection (PJI), at least, five intraoperative samples are taken before debridement and prosthesis removal in order to identify the causative organism. For the purpose of this study three additional intraoperative samples will be performed after debridement and antibiotic initiation and prior prosthesis implantation.
Description of outcomes of perioperative sample culture after surgical excision according to the identified germ in culture before excision. | 18 months
  In routine care procedure for prosthetic joint infection (PJI), at least, five intraoperative samples are taken before debridement and prosthesis removal in order to identify the causative organism. For the purpose of this study three additional intraoperative samples will be performed after debridement and antibiotic initiation and prior prosthesis implantation.
Description of outcomes of perioperative sample culture after surgical excision according to antibiotherapy duration from initiation until perioperative samples. | 18 months
  In routine care procedure for prosthetic joint infection (PJI), at least, five intraoperative samples are taken before debridement and prosthesis removal in order to identify the causative organism. For the purpose of this study three additional intraoperative samples will be performed after debridement and antibiotic initiation and prior prosthesis implantation.
Description of outcomes of perioperative sample culture prior surgical excision in patients treated with preoperative antibiotherapy. | 18 months
  In routine care procedure for prosthetic joint infection (PJI), at least, five intraoperative samples are taken before debridement and prosthesis removal in order to identify the causative organism. For the purpose of this study three additional intraoperative samples will be performed after debridement and antibiotic initiation and prior prosthesis implantation.
Description of outcomes of perioperative sample culture according to symptoms duration prior surgery. | 18 months
  In routine care procedure for prosthetic joint infection (PJI), at least, five intraoperative samples are taken before debridement and prosthesis removal in order to identify the causative organism. For the purpose of this study three additional intraoperative samples will be performed after debridement and antibiotic initiation and prior prosthesis implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Simon MARMOR, Doctorate, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No